CLINICAL TRIAL: NCT01330979
Title: A Phase 2 Open Label Study Assessing the Safety and Ocular Hypotensive Efficacy of AR-12286 in Patients With Open-angle Glaucoma or Ocular Hypertension
Brief Title: 24-hour Efficacy of AR-12286
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR-12286-CS204
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — AR-12286; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AR-12286 0.5% Ophthalmic Solution — Ophthalmic Solution

SUMMARY:
An open-label, non-comparative, pilot evaluation of the 24-hour ocular hypotensive efficacy of AR-12286 in patients with open-angle glaucoma or ocular hypertension

ELIGIBILITY:
* Inclusion criteria

  1. 40 to 80 years of age.
  2. Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT).
  3. Corrected visual acuity in each eye +1.0 logMAR or better by ETDRS in each eye (equivalent to 20/200).
  4. Able and willing to give signed informed consent and follow study instructions including two nights in UCSD sleep lab for physiological measurements.
* Exclusion criteria

Excluded from the study will be individuals with the following characteristics:

Ophthalmic (in either eye):

1. Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure or narrow irridocorneal angle. Note: Previous laser peripheral iridotomy is acceptable.
2. Intraocular pressure > 36 mm Hg.
3. Known hypersensitivity to any component of the formulation (benzalkonium chloride, etc.), or to topical anesthetics.
4. Previous glaucoma intraocular surgery or glaucoma laser procedures in study eye(s).
5. Refractive surgery in study eye(s) (e.g., radial keratotomy, PRK, LASIK, etc.).
6. Ocular trauma within the past six months, or ocular surgery or laser treatment within the past three months.
7. History or evidence of ocular infection, inflammation, clinically significant blepharitis or conjunctivitis at baseline (Visit 1), or of herpes simplex keratitis
8. Contact lens wear within 30 minutes of instillation of study medication.
9. Ocular medication of any kind within 30 days of Visit 1, with the exception of a) ocular hypotensive medications (which must be washed out according to the provided schedule), b) lid scrubs (which may be used prior to, but not after Visit 1) or c) lubricating drops for dry eye (which may be used throughout the study).
10. Clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe (i.e., cup-disc ratio > 0.8).
11. Central corneal thickness greater than 600 µ.
12. Any abnormality preventing reliable applanation tonometry of either eye.

    Systemic:
13. Clinically significant abnormalities in laboratory tests at screening.
14. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
15. Current use of cigarettes.
16. Irregular sleep schedule.
17. Participation in any investigational study within the past 30 days.
18. Changes of systemic medication that could have a substantial effect on IOP within 30 days prior to screening, or anticipated during the study.
19. Due to status of preclinical safety program, women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must not intend to become pregnant during the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | Day 28
  Intraocular pressure compared to baseline

SECONDARY OUTCOMES:
Intraocular pressure | Day 28
  Diurnal IOP

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, California, United States